CLINICAL TRIAL: NCT06268327
Title: Adding Adjuvant Cisplatin and Gemicitabine Versus Capecitabine in Triple-negative Breast Cancer Patients in Non pCR After Neoadjuvant Standard Chemotherapy
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sohaila Essam Mohamed, Assiut university Hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Adjuvant treatment in BC
Record Dates: First submitted 2023-11-19; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cisplatin; Gemcitabine; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cisplatin and gemicitabine (Experimental): patients with triple negative breast cancer will recieve adjuvant cisplatin and gemicitabine in non pathological complete response after neo-adjuvant standard chemotherapy with dose of cisplatin 70mg/m2 at day one and gemicitabine 1000mg/m2 day one and day eight every 21 day for six cycle
  Interventions: Drug: Cisplatin injection and gemcitabine
- capecitabine (Experimental): patients with triple negative breast cancer will recieve adjuvant capecitabin in non pathological complete response after neo-adjuvant standard chemotherapy with dose of capecitabine 1000-1250 mg/m2 every 21 day for six cycle
  Interventions: Drug: Capecitabine tablets

INTERVENTIONS:
Drug: Cisplatin injection and gemcitabine — Patients with operable, primary invasive noninflammatory early TNBC of stage I-IIIB and pathologically verified residual cancer cells (no pathological complete response) after neoadjuvant chemotherapy then underwent adjuvant treatment with gemcitabine plus cisplatin Pt will be followed up every 3 month in first year then every 6 month in the second year then followed up yearly Study will be conducted at Assiut University Hospital with sample size calculation BRACA will be done
  Arms: cisplatin and gemicitabine
Drug: Capecitabine tablets — Patients with operable, primary invasive noninflammatory early TNBC of stage I-IIIB and pathologically verified residual cancer cells (no pathological complete response) after neoadjuvant chemotherapy then underwent adjuvant treatment with capecitabine Pt will be followed up every 3 month in first year then every 6 month in the second year then followed up yearly Study will be conducted at Assiut University Hospital with sample size calculation BRACA will be done
  Arms: capecitabine

SUMMARY:
In our study; investigator aim To show efficacy and toxicity of Adjuvant cisplatin and gemcitabine in triple-negative breast cancer patients with non pathologically complete response after neoadjuvant chemotherapy To compare outcome of adjuvant cisplatin and gemcitabine versus capecitabine

DETAILED DESCRIPTION:
Patients with operable, primary invasive non inflammatory early TNBC of stage I-IIIB and pathologically verified residual cancer cells (no pathological complete response) after neoadjuvant chemotherapy then underwent adjuvant treatment with gemcitabine plus cisplatin Patients will be followed up every 3 month in first year then every 6 month in the second year then followed up yearly Study will be conducted at Assiut University Hospital with sample size calculation BRACA will be done

ELIGIBILITY:
Inclusion Criteria:

* Age: 20 years and older.
* Patients with no clinical/radiologic distant metastasis.
* Tumor type: Invasive ductal carcinoma or invaive lobular carcinoma.
* Tumor subtype: triple negative
* patients had operable, primary invasive, noninflammatory early stage I-IIIB TNBC (ER and PR <1%, HER2 score: 0 or 1)
* Patients with a good performance status (0/1)
* Patients with adequate hematological, cardiac, renal, and hepatic function

Exclusion Criteria:

* Patients who achieve pathologic complete response after neoadjuvant chemotherapy
* inflammatory breast cancer
* Breast cancer patients with distant metastasis
* Patient with hormonal receptor positive /HER2 +ve

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Adding adjuvant cisplatin and gemcitabine versus capecitabine in triple-negative Breast cancer patients with non pathologically complete response after neoadjuvant standard chemotherapy | 2 years
  2 years disease free survival which is calculated since time of surgery till occurance of local or distant recurrence

SECONDARY OUTCOMES:
Comparison of patients who receive cisplatin and gemcitabine versus capecitabine in Triple negative breast cancer | 3 years
  Compare if the investigated regimen is superior or same as standard regimen and the investigators will notice and document toxicity of both regimens including gastrointestinal toxicity, neurological toxicity, hematologic toxicity renal toxicity, ototoxicity and skin toxicity according to CTCAE version 4.1 also over all survival will be measured which is calculated from time of diagnosis till death or finishing our study minimum 3 years